CLINICAL TRIAL: NCT07353931
Title: A Master Protocol for Phase 3 Randomized, Double-Blind, Placebo-Controlled Studies to Investigate the Efficacy and Safety of Once Weekly Eloralintide in Adult Participants With Osteoarthritis Knee Pain, and Obesity or Overweight (ENLIGHTEN-4)
Brief Title: Efficacy and Safety of Eloralintide (LY3841136) in Participants With Osteoarthritis Knee Pain and Obesity or Overweight
Acronym: ENLIGHTEN-4
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27761; 2025-523768-19-00 (EU CTIS Number); J3R-MC-YDAN (Other: Eli Lilly and Company); J3R-MC-YOA1 (Other: Eli Lilly and Company); J3R-MC-YOA2 (Other: Eli Lilly and Company)
Record Dates: First submitted 2026-01-16; First posted 2026-01-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis; Overweight or Obesity
MeSH Terms: conditions — Osteoarthritis; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Eloralintide (YOA1) (Experimental): Participants will receive eloralintide subcutaneously (SC)
  Interventions: Drug: Eloralintide
- Placebo (YOA1) (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo
- Eloralintide (YOA2) (Experimental): Participants will receive eloralintide SC
  Interventions: Drug: Eloralintide
- Placebo (YOA2) (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eloralintide — Administered SC
  Other Names: LY3841136
  Arms: Eloralintide (YOA1); Eloralintide (YOA2)
Drug: Placebo — Placebo administered SC
  Arms: Placebo (YOA1); Placebo (YOA2)

SUMMARY:
The YDAN master protocol will support two independent studies, J3R-MC-YOA1 and J3R-MC-YOA2. Each study will investigate how well and safely Eloralintide (LY3841136) works in adults with obesity or overweight who have osteoarthritis (OA) of the knee with pain. Participation in the study will last about 75 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of 27 kilograms per square meter (kg/m²) or higher at screening
* Have a stable body weight (less than 5% body weight change) for 90 days prior to screening
* Have tried at least once to lose weight through diet but were unsuccessful
* Have osteoarthritis of the knee and at least one of the following conditions:

  * Be over 50 years old
  * Have morning knee stiffness that lasts about 30 minutes
  * Have a crackling or grinding sound or feeling in the knee

Exclusion Criteria:

* Have a prior or planned surgical treatment for obesity (liposuction, cryolipolysis, or abdominoplasty allowed if performed greater than 1 year before screening)
* Have a prior or planned endoscopic procedure and/or device-based therapy for obesity (prior device-based therapy acceptable if device removal was more than 6 months prior to screening)
* Have type 1 diabetes, type 2 diabetes, or any other type of diabetes
* Have an active knee infection
* Have had within 90 days prior to screening:

  * heart attack
  * stroke
  * coronary artery revascularization
  * unstable angina, or
  * hospitalization due to congestive heart failure
* Have a history or diagnosis of New York Heart Association Functional Classification Class IV congestive heart failure
* Have taken medications or alternative remedies intended for weight loss within 90 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 64
  Percent Change from Baseline in Body Weight
Change from Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score | Baseline, Week 64
  Change from Baseline in the WOMAC Pain Subscale Score

SECONDARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 64
  Change from Baseline in SBP
Percent Change from Baseline in Triglycerides | Baseline, Week 64
  Percent Change in Baseline in Triglycerides
Change from Baseline in Short Form-36 (SF-36 v2) Acute Form Physical Functioning Domain Score | Baseline, Week 64
  Change from Baseline in SF-36 v2 Score
Percent Change from Baseline in High Sensitivity, C-reactive Protein (hsCRP) | Baseline, Week 64
  Percent Change from Baseline in hsCRP
Change from Baseline in the WOMAC Physical Function Subscale Score | Baseline, Week 40, Week 64
  Change from Baseline in the WOMAC Physical Function Subscale Score
Change from Baseline WOMAC Pain Subscale Score | Baseline, Week 40
  Change from Baseline WOMAC Pain Subscale Score
Change from Baseline in Distance Walked During the 6-Minute Walk Test | Baseline, Week 64
  Change from Baseline in Distance Walked During the 6-Minute Walk Test
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 64
  Change from Baseline in BMI
Change in Medication Use | Baseline, Week 64
  Change in Medication Use
Change from Baseline in SF-36v2 Acute Form Domain Scores With Exception of the Physical Functioning Domain Score | Baseline, Week 64
  Change from Baseline in SF-36v2 Acute Form Domain Scores With Exception of the Physical Functioning Domain Score
Change from Baseline in Health Status EQ-5D-5L Health State Utility | Baseline, Week 64
  Change from Baseline in Health Status EQ-5D-5L Health State Utility
Percent Change from Baseline in Fasting Insulin | Baseline, Week 64
  Percent Change from Baseline in Fasting Insulin
Percent Change from Baseline in Total Cholesterol | Baseline, Week 64
  Percent Change from Baseline in Total Cholesterol
Change from Baseline in Waist Circumference | Baseline, Week 64
  Change from Baseline in Waist Circumference
Percent Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 64
  Percent Change from Baseline in HbA1c
Change from Baseline in WOMAC Stiffness Subscale Score | Baseline, Week 64
  Change from Baseline in WOMAC Stiffness Subscale Score
Change from Baseline in WOMAC Total Score | Baseline, Week 64
  Change from Baseline in WOMAC Total Score
Achievement of Improved Categorical Shift in Patient Global Impression of Severity (PGIS) - Target Knee Pain | Baseline, Week 64
  Achievement of Improved Categorical Shift in PGIS - Target Knee Pain
Achievement of Improved Categorical Shift in Patient Global Impression of Severity (PGIS) - Target Knee Function | Baseline, Week 64
  Achievement of Improved Categorical Shift in PGIS - Target Knee Function
Change from Baseline in Average Pain Intensity Numeric Rating Scale (API-NRS) Score | Baseline, Week 64
  Change from Baseline in API-NRS Score
Change from Baseline in Worst Pain Intensity Numeric Rating Scale (WPI-NRS) Score | Baseline, Week 64
  Change from Baseline in WPI-NRS Score
Pharmacokinetics (PK): Maximum Concentration at Steady State (Cmax, ss) | Baseline through Week 64
  PK: Cmax, ss
PK: Area Under the Concentration Versus Time Curve for One Dosing Interval at Steady State (AUC(0-T)ss) | Baseline through Week 64
  PK: AUC(0-T)ss
Number of Participants with Allowed Concomitant Pain Medication | Baseline, Week 64
  Number of Participants with Allowed Concomitant Pain Medication

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (155):
- United States (35):
  - AMR Clinical, Mobile, Alabama
  - Care Access - 801 South Power Road, Mesa, Mesa, Arizona
  - Elite Pain and Spine Institute - South Crimson Road, Mesa, Arizona
  - Tucson Orthopaedic Institute - North Wyatt Drive, Tucson, Arizona
  - Ark Clinical Research - Fountain Valley, Fountain Valley, California
  - Wolverine Clinical Trials, Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Care Access - St. Petersburg, St. Petersburg, Florida
  - Conquest Research, Winter Park, Florida
  - Orita Clinical Research, Decatur, Georgia
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Qualmedica Research, LLC, Evansville, Indiana
  - AMR Clinical, Newton, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Skylight Health Research - Burlington, Burlington, Massachusetts
  - Care Access - Quincy, Quincy, Massachusetts
  - Ellipsis Research Group - Brooklyn - 7th Street, Brooklyn, New York
  - Rochester Clinical Research - Buffalo, Buffalo, New York
  - NYC Research INC, Long Island City, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - AMC Research, LLC, Matthews, North Carolina
  - Central States Research, Tulsa, Oklahoma
  - Heritage Valley Multispecialty Group, Inc, Beaver, Pennsylvania
  - Keystone Clinical Studies, Plymouth Meeting, Pennsylvania
  - JCCT - Juno Bellaire Site, Bellaire, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - Valley Institute of Research - Fort Worth, Fort Worth, Texas
  - Care Access - Houston, Houston, Texas
  - VIP Trials, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - AMR Clinical, South Jordan, Utah
- Argentina (15):
  - Centro Privado de Medicina Familiar / Mindout Research, Buenos Aires
  - Organizacion Medica de Investigacion, Buenos Aires
  - Stat Research S.A., Buenos Aires
  - CIPREC, Buenos Aires
  - Centro Médico Arsema, Buenos Aires
  - APRILLUS Asistencia E Investigacion, CABA
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - INECO Neurociencias Oroño, Rosario
  - Instituto Especialidades de la Salud Rosario, Rosario
  - Medicina Reumatológica, San Fernando
  - Instituto de Alta Complejidad San Isidro, San Isidro
  - Centro Polivalente de Asistencia e Investigacion Clinica - CER San Juan, San Juan
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán
  - Go Centro Medico San Nicolás, San Nicolás
- Belgium (8):
  - Antwerp University Hospital, Edegem
  - Reuma Clinic, Locatie Jaarbeurslaan, Genk
  - UZ Gent, Ghent
  - Kormont, Kluisbergen
  - UZ Leuven, Leuven
  - Meclinas, Mechelen
  - ZNA Jan Palfijn, Merksem
  - Medisch Centrum Latem (Hip Clinic) - Algemeen Ziekenhuis Maria Middelares Location, Sint-Martens-Latem
- Brazil (6):
  - Centro de Pesquisa Sao Lucas, Campinas
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - CPHosp Medicina, Ensino e Pesquisa (CPQuali), São Paulo
  - INTEGRA - Pesquisa Clínica e Infusões, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
- Canada (7):
  - Apex Trials, Guelph
  - G.R.M.O. (Groupe de recherche en maladies osseuses) Inc., Québec
  - Diex Recherche Inc. Division Quebec, Québec
  - Stouffville Medical Research Institute Inc., Stouffville
  - Maple Leaf Research, Toronto
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto
  - Diex Recherche Inc. Division Victoriaville, Victoriaville
- China (19):
  - Beijing Ji Shui Tan Hospital, Beijing
  - The First Afflilated Hospital of Bengbu Medical College, Bengbu
  - Jilin Province People's Hospital, Changchun
  - Xiangya Hospital Central South University, Changsha
  - 2nd Affiliated Hospital Chongqing Medical Universi, Chongqing
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated hospital of Zhejiang University school of medicine, Hangzhou
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang
  - Nanjing First Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - The first affiliated hospital of Ningbo university, Ningbo
  - Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital,Fudan University, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Hospital, Tianjin
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan
- Czechia (5):
  - Pratia Brno, Brno
  - Revmatologie.s.r.o., Brno
  - INREA s.r.o., Ostrava
  - Pratia Pardubice a.s., Pardubice
  - Medical Plus Research, Uherské Hradiště
- Denmark (3):
  - Sanos Clinic - Nordjylland, Gandrup
  - Sanos Clinic, Herlev
  - Sanos Clinic - Syddanmark, Vejle
- Germany (8):
  - Siteworks GmbH - Bochum, Bochum
  - Private Practice - Dr. Kai Könemann & Dr. Henrik Könemann, Bünde
  - StudyPoint Duisburg, Duisburg
  - HRF II - Hamburger Rheuma Forschungszentrum II MVZ für Rheumatologie und Autoimmunmedizin Hamburg GmbH / -T, Hamburg
  - Siteworks - Karlsruhe, Karlsruhe
  - AmBeNet GmbH, Leipzig
  - CDG Studienambulanz Hartard, München
  - Dedicated Research Site FutureMeds, Offenbach
- Japan (15):
  - National Hospital Organization Chiba Medical Center, Chiba
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Tokyo Asbo Clinic, Chūōku
  - Shin Komonji Hospital, Kitakyushu-Shi
  - Goto Orthopedic Surgery Clinic, Miyazaki
  - Komagidai Clinic, Nagareyama
  - Fujigaki Clinic, Ōita
  - Saitama City Hospital, Saitama
  - Ibaraki Seinan Medical Center Hospital, Sashima
  - Ogura Orthopedics Surgery, Sendai
  - Katsura Garden Orthopedics, Sendai
  - Ooimachi Orthopedic Surgery and surgery Clinic, Shinagawa-ku Tokyo
  - Masumoto Orthopedics Clinic, Suginami City
  - National Hospital Organization Toyohashi Medical Center, Toyohashi
  - Yamagata Tokushukai Hospital, Yamagata
- Mexico (9):
  - Investigacion y Biomedicina de Chihuahua, Chihuahua City
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, S.C., Ciudad Madero
  - Diseno y Planeacion en Investigacion Medica - Guadalajara - Calle Amado Nervo, Guadalajara
  - Unidad de Investigación Clínica y Atención Médica HEPA S.C., Guadalajara
  - RM Pharma Specialists - Unidad Especializada en Datos, Mexico City
  - Kohler & Milstein Research S.A. De C.V., Mérida
  - IMED Internal Medicine Clin Trials, Monterrey
  - UBAM Unidad Biomedica Avanzada Monterrey, Monterrey
  - Centro de investigación y control metabólico, Monterrey
- Puerto Rico (2):
  - Dorado Medical Complex, Dorado
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
- South Korea (8):
  - Keimyung University Dongsan Hospital, Daegu
  - Boramae Medical Center, Dongjak-gu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - The Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si
- Taiwan (7):
  - Changhua Christian Hospital, Changhua County
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- United Kingdom (8):
  - Velocity Clinical Research, Bristol, Bristol
  - FutureMeds Glasgow - CPS Research, Glasgow
  - FutureMeds - London, London
  - Futuremeds-Newcastle, Newcastle
  - Atlantic Medical, Penzance
  - Woodstock Bower Surgery, Rotherham
  - Panthera Biopartners - Sheffield, Sheffield
  - Panthera Clinic - York, York

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Lilly Trials — https://trials.lilly.com/en-US/trial/660855